CLINICAL TRIAL: NCT06056583
Title: Postpartum Activity and Expression of BCRP and OCT1 Drug Transporters in the Mammary Gland
Brief Title: Drug Excretion in Breast Milk
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mary Hebert, Professor: Pharmacy; Adjunct Professor, Obstetrics & Gynecology, University of Washington
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00018397; R01HD112282 (NIH)
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Postpartum; Lactation; Drugs in Breast Milk; Mammary Drug Transporters; BCRP; OCT1
Keywords: breast milk; lactation; cimetidine; proteomics; OCT1; BCRP; OCTN2; PEPT2; ENT1; CNT3; MRP1; OATP2B1; OATP3A1; OCT2; postpartum; pharmacokinetics
MeSH Terms: conditions — Breast Feeding | interventions — Cimetidine

STUDY DESIGN:
Intervention Model Description: This is a phase 1 study design of an approved drug to evaluate the time-course for the expression and activity of OCT1 and BCRP in the mammary gland 3-5 weeks, 3-4 months and 6-8 months postpartum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Lactating Women (Other): Healthy Lactating Women will be studied on 3 study days and serve as their own control.
  Interventions: Drug: Cimetidine 200 MG

INTERVENTIONS:
Drug: Cimetidine 200 MG — Cimetidine will serve as the probe drug
  Other Names: Tagamet

SUMMARY:
This is a prospective, non-randomized, phase I study design evaluating the in vivo activities and expression of OCT1 and BCRP in mammary gland of lactating women at three time points postpartum.

DETAILED DESCRIPTION:
Each woman will receive a single oral dose of cimetidine 200 mg on each of 3 study days (3-5 weeks, 3-4 months, and 6-8 months postpartum) followed by serial collection of blood, urine and breast milk samples over 12-hours. Cimetidine concentrations will be assay using a validated LC/MS/MS assay. Subjects will be genotyped for OCT1 and BCRP. Mammary epithelial cells will be isolated from breast milk and transporter expression will be quantified. Each woman will serve as her own control.

ELIGIBILITY:
Inclusion criteria

1. Healthy postpartum women
2. 18-50 years of age and their infants
3. Able to provide written informed consent

Exclusion criteria

1. Receiving cimetidine within the 3 days prior to each study day. Concomitant administration of cimetidine will confound interpretation of study results.
2. Hypersensitivity to cimetidine Patients with known allergic reactions to cimetidine will be excluded for safety reasons
3. Receiving medication known to interact with cimetidine: OCT, BCRP, CYP3A4, CYP2D6, CYP1A2 and CYP2C9 substrates (e.g. amiodarone, clopidogrel, diazepam, ketoconazole, metformin, nifedipine, phenytoin, procainamide, theophylline,tricyclic antidepressants and warfarin) Patients with drug interactions will be excluded for safety reasons.
4. Receiving BCRP inhibitors/inducers (afatinib, aripipraxole, axitinib, cimetidine, cyclosporine, curcumin/tumeric, delavirdine, efavirenz, elacridar, elvitegravir, etravirine, FTC, 5-fluorouracil, fluvastatin, imatinib, lanzoprazole, lapatinib, lopinavir, maraviroc, nelfinavir, nebicapone, nilotinib, novobiocin, oltipraz, omeprazole, pantoprazole, phenobarbital, promazine, rabeprazole, riboflavin, rifampicin, risperidone, saquinavir, sirolimus, sorafenib, sulfasalazine, sunitinib, tacrolimus, tariquidar, telaprevir, telatinib, teriflunomide, tolcapone, triflunomide, trametinib, trifluoperazine, venlafaxine, zidonuvir), OCT1 inhibitors/inducers (acyclovir, amantadine, amiloride, amitriptyline, bucindolol, carvedilol, chlorpheniramine, chlorpromazine, cimetidine, citalopram, clonidine, clopidogrel, clotrimazole, clozapine, cocaine, corticosterone, cyclosporine, daclatasvir, darunavir, desipramine, dextromethorphan, diltiazem, disopyramide, dronedarone, efavirenz, famotidine, fentanyl, fluvoxamine, formoterol, fuloxetine, griseofulvin, doxazosine, ganciclovir, guanfacine, imipramine, indinavir, isavuconazole, itraconazole, ketoconazole, lamotrigine, lasmiditan, levofloxacin, levomepromazine, lidocaine, maprotiline, methylnicotinamide, morphine, moxifloxacin, nefazodone, nelfinavir, nevirapine, nicotine, nomifensine, ondansetron, oxybutynin, paroxetine, pentamidine, phenoxybenzamine, prazosin, probenecid, procainamide, propafenone, pyrazinamide, quetiapine,quinidine, quinine, reboxetine, remoxidpride, reseripine, rifampicin, ritonavir, salmeterol, saquinavir, tramadol, trimethoprim, trimipramine, verapamil) Inhibitors and inducers of the drug transporters will confound data analysis and interpretation.
5. Kidney disease could confound data analysis and interpretation. Therefore, patients with known kidney disease with documented renal function impairment will be excluded from the study. Current serum creatinine > 1.2 mg/dL in their medical record will be excluded.
6. Known liver disease Liver disease will confound data analysis and interpretation. Therefore, patients with known significant liver disease will be excluded from the study. Current ALT exceeding 2-times the upper limit of normal in their medical record will be excluded.
7. Inability to fast for 4 hours prior to the study. To limit PK variability across study days, subjects will be requested to fast for 4 hours prior to each study day.
8. Smokers (tobacco or other nicotine containing products Nicotine interacts with OCT1 and will confound data analysis and interpretation

Ages: 14 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Mammary clearance of cimetidine | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Cimetidine excretion into breast milk at three postpartum stages
Mammary epithelial cell expression of BCRP | 3-5 weeks, 3-4 months and 6-8 months postpartum
  BCRP protein expression in MECs at three postpartum stages
Mammary epithelial cell expression of OCT1 | 3-5 weeks, 3-4 months and 6-8 months postpartum
  OCT1 protein expression in MECs at three postpartum stages

SECONDARY OUTCOMES:
Cimetidine relative infant dose and infant concentration | 3-5 weeks, 3-4 months and 6-8 months postpartum
  cimetidine relative infant dose (RID) and infant concentration
Relationship between OCT1 expression and activity | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effect of time postpartum on OCT1 protein expression in MECs and correlation with cimetidine mammary CL
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine CL/F
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine renal CL
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine renal secretion CL
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine mammary CL
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine AUC
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine Cmax
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine Tmax
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine half-life
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine apparent oral volume of distribution
Maternal cimetidine PK | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effects of time postpartum on cimetidine elimination rate constant
Relationship between BCRP expression and activity | 3-5 weeks, 3-4 months and 6-8 months postpartum
  Effect of time postpartum on BCRP protein expression in MECs and correlation with cimetidine mammary CL

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hebert, PharmD, FCCP, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We are committed to share data with the academic community and researcher-at-large. We will adhere to the NIH Grant Policy on Sharing Research Data and Resources. That is, after final data collection and analysis and after full peer review is performed on our data, the de-identified data generated by this project will be made available when requested by the academic community and researchers-at-large contingent upon Material Transfer Agreements with the University of Washington.
Supporting Information: CSR
Time Frame: After peer review and publication of data.
Access Criteria: We are committed to share data with the academic community and researcher-at-large. We will adhere to the NIH Grant Policy on Sharing Research Data and Resources. That is, after final data collection and analysis and after full peer review is performed on our data, the de-identified data generated by this project will be made available when requested by the academic community and researchers-at-large contingent upon Material Transfer Agreements with the University of Washington.